CLINICAL TRIAL: NCT06577441
Title: A Randomized Phase II Trial of Enasidenib-Based Therapies Versus Cedazuridine-Decitabine in Higher-Risk IDH2-Mutated Myelodysplastic Syndrome: A MyeloMATCH Sub-Study
Brief Title: Testing the Addition of an IDH2 Inhibitor, Enasidenib, to Usual Treatment (Cedazuridine-Decitabine) for Higher-Risk Myelodysplastic Syndrome (MDS) With IDH2 Mutation (A MyeloMATCH Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-07049; NCI-2024-07049 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MM1MDS-A01 (Other: Alliance for Clinical Trials in Oncology); MM1MDS-A01 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2024-08-28; First posted 2024-08-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Specimen Handling; Biopsy; decitabine and cedazuridine drug combination; enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regimen 1 (ASTX727) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR, CRL, or CRh at the end of cycle 6 may cross-over to Regimen 2. Patients who experience CR, PR, or SD any time after 4 cycles of treatment may be reassessed in order to go to a higher myeloMATCH tier assignment or to TAP. Patients also undergo bone marrow biopsy and aspiration throughout the study. Patients may also undergo optional buccal swab on study, and/or optional additional bone marrow aspiration and blood sample collection on study and at disease progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine
- Regimen 2 (ASTX727, enasidenib) (Experimental): Patients receive ASTX727 PO QD on days 1-5 and enasidenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience CR, PR, or SD any time after 4 cycles of treatment may be reassessed in order to go to a higher myeloMATCH tier assignment or to TAP. Patients also undergo bone marrow biopsy and aspiration throughout the study. Patients may also undergo optional buccal swab on study, and/or optional additional bone marrow aspiration and blood sample collection on study and at disease progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Enasidenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo buccal swab and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Drug: Enasidenib — Given PO
  Other Names: AG 221; AG-221; AG221; CC-90007 Free Base
  Arms: Regimen 2 (ASTX727, enasidenib)

SUMMARY:
This phase II MyeloMATCH treatment trial compares the usual treatment of cedazuridine-decitabine (ASTX727) to the combination treatment of ASTX727 and enasidenib in treating patients with higher-risk, IDH2-mutated myelodysplastic syndrome (MDS). ASTX727 is a combination of two drugs, decitabine and cedazuridine. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Enasidenib is an enzyme inhibitor that may stop the growth of cells by blocking some of the enzymes needed for cell growth. Giving ASTX727 in combination with enasidenib may be effective in treating patients with higher-risk IDH2-mutated MDS.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the complete remission (CR) rate of enasidenib + decitabine and cedazuridine (ASTX727) and ASTX727 monotherapy in patients with higher-risk IDH2-mutated MDS using International Working Group 2023 (IWG2023) response criteria.

SECONDARY OBJECTIVES:

I. To estimate the median event-free survival (EFS) at designated time point(s) for each treatment arm.

II. To estimate the median overall survival (OS) at designated time point(s) for each treatment arm.

III. To estimate the frequency and severity of toxicities with each regimen in this patient population.

IV. To estimate the median time to response for each treatment arm. V. To estimate the median duration of response for each treatment arm. VI. To estimate the IDH2 variant allele frequency (VAF) reduction for each treatment arm.

VII. To estimate the rate of allogeneic hematopoietic cell transplantation for each treatment arm.

VIII. To compare rates of partial response (PR), CR with limited count recovery (CRL), CR with partial count recovery (CRh), and hematologic improvement (HI) using IWG 2023 response criteria between treatment arms.

IX. To compare the measurable residual disease (MRD) kinetics by flow cytometry and next generation sequencing (NGS) at designated time point(s) at the end of cycle 4 & 6 and to assess any correlation with clinical outcomes (e.g. CR, EFS, OS).

X. To estimate the median time to transformation of MDS to acute myeloid leukemia (AML).

EXPLORATORY OBJECTIVES:

I. To estimate CR rate, median EFS, and median OS in patients treated with ASTX727 monotherapy that crossover to the treatment arm with ASTX727 + enasidenib after 6 cycles if CR is not achieved.

II. To estimate CR rate, median EFS, and median OS for patients based on Molecular International Prognostic Scoring System (IPSS-M) prognostic risk score at diagnosis, stratified for score level.

III. To estimate concordance between centrally-performed molecular studies and cytogenetics to those done locally.

OUTLINE: Patients are randomized to 1 of 2 regimens.

REGIMEN 1: Patients receive ASTX727 orally (PO) once daily (QD) on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR, CRL, or CRh at the end of cycle 6 may cross-over to Regimen 2. Patients who experience CR, PR, or stable disease (SD) any time after 4 cycles of treatment may be reassessed in order to go to a higher myeloMATCH tier assignment or to Tier Advancement Pathway (TAP). Patients also undergo bone marrow biopsy and aspiration throughout the study. Patients may also undergo optional buccal swab on study, and/or optional additional bone marrow aspiration and blood sample collection on study and at disease progression.

REGIMEN 2: Patients receive ASTX727 PO QD on days 1-5 and enasidenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience CR, PR, or SD any time after 4 cycles of treatment may be reassessed in order to go to a higher myeloMATCH tier assignment or to TAP. Patients also undergo bone marrow biopsy and aspiration throughout the study. Patients may also undergo optional buccal swab on study, and/or optional additional bone marrow aspiration and blood sample collection on study and at disease progression.

After completion of study treatment, patients are followed up every 6 months for up to 5 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* GENERAL MYLEOMATCH REGISTRATION CRITERIA:

  * Patients must be registered to the Master Screening and Reassessment Protocol (MSRP) and assigned to this protocol by the MATCHBox Treatment Verification Team.
  * Participants must not have received prior anti-cancer therapy for AML or MDS.

    * Note: Hydroxyurea to control the white blood cell count (WBC) is allowed.
    * Note: Prior erythroid stimulating agent (ESA) is not considered prior therapy for the purposes of eligibility.
  * Participants must not be currently receiving any cytarabine-containing therapy other than up to 1 g/m^2 of cytarabine, which is allowed for urgent cytoreduction. The use of prior hydroxyurea, all-trans retinoic acid (ATRA), BCR-ABL directed tyrosine kinase inhibitor, erythropoiesis-stimulating agent, thrombopoietin receptor agonist and lenalidomide is allowed
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients must have a morphologically-confirmed diagnosis of MDS with a Revised International Prognostic Scoring System (IPSS-R) score ≥ 4.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients must have a detectable pathogenic IDH2 mutation based on the National Cancer Institute (NCI) Myeloid Panel.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): No prior treatment with deoxyribonucleic acid (DNA) methyltransferase inhibitors (ASTX727, azacitidine, or decitabine).
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Prior treatment with growth factors (ESA, granulocyte colony-stimulating factor [g-CSF], thrombopoietin [TPO] agonist), lenalidomide or luspatercept is allowed with a maximum limit of 1 month of exposure.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients with therapy-related MDS are allowed.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Age ≥ 18 years.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Total bilirubin ≤ 1.5 x upper limit of normal (ULN)

  * Unless elevated due to Gilbert's syndrome. In patients with Gilbert's syndrome, if the total bilirubin is ≤ 3.0 x ULN, then they are eligible for enrollment.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) ≤ 3.0 x upper limit of normal (ULN).
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Creatinine clearance ≥ 30 mL/min

  * To be calculated using Cockroft Gault formula.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Not pregnant and not nursing, because this study involves: an agent that has known genotoxic, mutagenic and teratogenic effects.

  * Therefore, for women of childbearing potential only, a negative pregnancy test done as part of screening lab work prior to registration is required.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1): Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Patients on the ASTX727 monotherapy arm (Regimen 1) that do not achieve a CR (complete response), CRL (CR with limited count recovery), or CRh (CR with partial count recovery) after completing 6 cycles of study treatment.
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): ECOG performance status ≤ 2.
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Total bilirubin ≤ 1.5 x upper limit of normal (ULN).

  * Unless elevated due to Gilbert's syndrome. In patients with Gilbert's syndrome if the total bilirubin is ≤ 3.0 x ULN, then they are eligible for enrollment.
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): AST (SGOT)/ALT (SGPT) ≤ 3.0 x upper limit of normal (ULN)
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Creatinine clearance ≥ 30 mL/min

  * To be calculated using Cockroft Gault formula.
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2): Not pregnant and not nursing, because this study involves: an agent that has known genotoxic, mutagenic and teratogenic effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | Up to 4 cycles of treatment
  Will be assessed using the International Working Group 2023 (IWG2023) criteria. Will compare the CR rate between the two treatment arms to determine if patients treated with enasidenib + ASTX727 have a statistically significantly higher CR rate than patients treated with the ASTX727 monotherapy.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Time from randomization to either a failure to achieve a CR, CR with limited count recovery (CRL), or CR with partial count recovery (CRh) after four cycles of treatment, relapse, or death due to any cause, assessed up to 18 months
  Sensitivity analyses will be conducted. Will use the methods of Kaplan-Meier as well as Cox regression models.
Overall survival (OS) | Time from randomization to death due to any cause, assessed up to 18 months
  Will use the methods of Kaplan-Meier as well as Cox regression models.
Time to response | Time from randomization to documented response, assessed up to 5 years
  Will be assessed only among patients who achieve a response (CR, CRL, or CRh). Will utilize the methods of Kaplan-Meier as well as Cox regression models.
Duration of response | From patient first achieves a response until either progression or death, assessed up to 5 years
  Will be assessed only among patients who achieve a response (CR, CRL, or CRh). Will use the methods of Kaplan-Meier as well as Cox regression models.
Incidence of adverse events | Up to 4 weeks after completion of study treatment
  Will be determined using the Common Terminology Criteria for Adverse Events version 5 criteria. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. Will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The incidence of severe (grade 3+) adverse events or toxicities will be described for each treatment arm, but will also be compared between the arms. Fisher's exact tests will be used to quantitatively compare the incidence of severe as well as specific toxicities of interest and will graphically assess differences in maximum grades observed for toxicities.
Change in IDH2 variant allele frequency (VAF) | Baseline to end of cycle 4 and 6
  Will report the percent change of VAF along with a 95% confidence interval.
Allogeneic stem cell transplantation rate | Up to 5 years
  Will report along with a 95% confidence interval for each treatment arm.
Measurable residual disease rate | At the end of cycle 4 and 6
  Will be measured by flow cytometry and next generation sequencing. Will be compared and used to determine association with clinical outcomes such as CR, EFS, or OS.
Cytogenetic and molecular features | Up to 5 years
  Cytogenetic and molecular classifications including Molecular International Prognostic Scoring System will be compared and used to determined association with clinical outcomes such as CR, EFS, and OS.
Time to transformation of myelodysplastic syndrome to acute myeloid leukemia (AML) | From randomization to transformation to AML or death from any causes, assessed up to 5 years
  Will utilize the methods of Kaplan-Meier as well as Cox regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Anand A Patel, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (124):
- United States (122):
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Mills Health Center, San Mateo, California
  - Memorial Hospital West, Pembroke Pines, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm